CLINICAL TRIAL: NCT04209595
Title: Phase I/II Trial of PLX038 (PEGylated SN38) and Rucaparib in Solid Tumors and Small Cell Cancers
Brief Title: PLX038 (PEGylated SN38) and Rucaparib in Solid Tumors and Small Cell Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anish Thomas, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200013; 20-C-0013
Record Dates: First submitted 2019-12-21; First posted 2019-12-24 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Small Cell Lung Cancer; Extra-Pulmonary Small Cell Carcinomas
Keywords: PARP Inhibitor; Chemotherapy; DDR Inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — rucaparib; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I Arm 1 Level -1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 200 mg (Experimental): Phase I - Participants with solid tumors enrolled to PLX038 (PEGylated SN38) and rucaparib escalation dose levels.
  PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 200 mg by mouth (PO)
  Interventions: Drug: PLX038; Drug: Rucaparib; Drug: Ondansetron
- Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg (Experimental): Phase I - Participants with solid tumors enrolled to PLX038 (PEGylated SN38) and rucaparib escalation dose levels.
  PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 400 mg by mouth (PO)
  Interventions: Drug: PLX038; Drug: Rucaparib; Drug: Ondansetron
- Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg (Experimental): Phase I Participants with solid tumors enrolled to PLX038 (PEGylated SN38) and rucaparib escalation dose levels.
  PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 300 mg by mouth (PO)
  Interventions: Drug: PLX038; Drug: Rucaparib; Drug: Ondansetron
- Phase IIA Arm 2 (Experimental): Phase IIA Participants with small cell lung cancer (SCLC) enrolled at the maximum tolerated dose (MTD) of PLX038 (PEGylated SN38) and rucaparib after the MTD of PLX038 and rucaparib is established.
  Level 2, PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 3, PLX038, every 3 weeks, 1.7 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 4, PLX038, every 3 weeks, 2.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 2A PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 400 mg by mouth (PO); and/or Level 3A. PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 600 mg by mouth (PO).
  Interventions: Drug: PLX038; Drug: Rucaparib; Drug: Ondansetron
- Phase IIB Arm 2 (Experimental): Phase IIB Participants with extra-pulmonary small cell carcinomas enrolled at the maximum tolerated dose (MTD) of PLX038 (PEGylated SN38) and rucaparib after the MTD of PLX038 and rucaparib is established.
  Level 2, PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 3, PLX038, every 3 weeks, 1.7 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 4, PLX038, every 3 weeks, 2.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 2A PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 400 mg by mouth (PO); and/or Level 3A. PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 600 mg by mouth (PO).
  Interventions: Drug: PLX038; Drug: Rucaparib; Drug: Ondansetron

INTERVENTIONS:
Drug: PLX038 — Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. PLX038 (PEGylated SN38) will be administered as a 1 hour (-10 minutes / +30 minutes) intravenous (IV) infusion on Day 1 of each cycle (21 days).
  Other Names: PEGylated SN38
Drug: Rucaparib — Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. Rucaparib will be given orally at designated dose twice a day on days 5 to 19 of every 21-day cycle.
  Other Names: Rubraca
Drug: Ondansetron — Participants will be recommended to have 8 mg of ondansetron taken with a small meal or snack to prevent nausea and vomiting approximately 30 minutes prior to each dose of rucaparib.
  Other Names: Zofran

SUMMARY:
Background:

Drugs known as poly-adenosine diphosphate ribose polymerase (PARP) inhibitors are known to help stop tumor growth in patients with breast, ovarian cancers and many other cancers including prostate and pancreatic cancers. Many research studies done in animals and human cells have shown that these types of drugs can improve how well chemotherapy works. Standard chemotherapy can be too toxic to be combined with PARP inhibitors. In this study, we use a new form of chemotherapy called PLX038 (PEGylated SN38) to see if it can be safely combined with PARP inhibitors to shrink tumors.

Objective:

To find a safe combination of PLX038 and rucaparib, and to see if this mix will cause tumors to shrink.

Eligibility:

People age 18 and older with solid tumors, small cell lung cancer (SCLC), or small cell cancer outside their lungs.

Design:

Participants will be screened with:

Physical exam

Blood tests

Records of their diagnosis (or they will have a tumor biopsy).

A review of their symptoms and medications.

A review of their ability to perform their normal activities.

Electrocardiograms, to measure the electrical activity of the heart.

Computed tomography (CT) scans of the chest, abdomen, and pelvis. CT scans are a series of X-rays.

Participants will get PLX038 by intravenous catheter on Day 1 of each cycle (1 cycle = 21 days). For this, a small plastic tube is put into an arm vein. They will take rucaparib twice daily by mouth on Days 3 to 19 of each cycle. They will keep a medicine diary.

Participants may give a hair sample. They may have optional tumor biopsies.

Screening tests are repeated throughout the study.

About 30 days after treatment ends, participants will have a safety follow-up visit. They will give blood samples, talk about their health, and get a physical exam. Then they will be called or emailed every 6 months....

DETAILED DESCRIPTION:
Background:

* We hypothesize that a dose-escalation strategy that incorporates tumor targeted deoxyribonucleic acid (DNA)-damaging chemotherapy and DNA-damage response (DDR) inhibitors could allow safe and effective administration of DNA damage response (DDR) inhibitor-chemotherapy combination.
* PLX038 is a PEGylated conjugate of SN38 with improved properties including increased solubility, higher exposure and longer half-life. SN-38 is the active metabolite of CPT-11 (irinotecan) that inhibits topoisomerase 1 (Top1) and causes DNA strand breakage. As a specific DNA damaging agent, SN-38 enhances cell kill in tumors deficient in the DNA-damage response and when combined with inhibitors of the DDR.
* Rucaparib is a potent oral poly ADP ribose polymerase (PARP) inhibitor that is approved for the maintenance treatment of participants with recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in a complete or partial response to platinum-based chemotherapy.
* We hypothesize that the combination of PLX038 plus rucaparib is more efficacious than either agent alone.

Objectives:

* Phase I: To identify the maximum tolerated dose (MTD) of PLX038 in combination with rucaparib.
* Phase II: To assess the efficacy with respect to clinical benefit rate (CBR) (CR+PR+SD) for 4 months according to Response Evaluation Criteria (RECIST 1.1) of a combination of PLX038 and rucaparib in participants with small cell lung cancer and extra-pulmonary small cell carcinomas.

Eligibility:

* Subjects with histologically confirmed solid tumors (Phase I) OR histologically or cytologically confirmed small cell lung cancer (SCLC) (Phase II) OR histologically or cytologically confirmed extra-pulmonary small cell carcinomas (Phase II).
* Age greater than or equal to 18 years
* Subjects must have evaluable, or measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate organ function

Design:

* This is an open label Phase I/II trial accruing initially one cohort to determine maximum tolerated dose (MTD) of combined treatment of PLX038 and rucaparib (Phase I); and to examine the safety and efficacy of PLX038 in combination with rucaparib in the following cohort (Phase II).
* PLX038 will be administered by intravenous (IV) infusion on day 1 of every 21-days cycle, rucaparib will be administered by mouth (PO) twice daily on days 6 to 19 of every cycle.
* Treatment will continue until progression or unacceptable toxicity.
* Biomarkers of participant response to treatment will be investigated in an exploratory manner pre- and post-treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects with:

  * histologically confirmed solid tumors (Phase I), OR
  * histologically or cytologically confirmed small cell lung cancer (SCLC) (Phase II), OR
  * histologically or cytologically confirmed extra-pulmonary small cell carcinomas (Phase II).
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of PLX038 (PEGylated SN38) in combination with rucaparib in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Subjects must have progressed on or after standard first-line systemic chemotherapy and have no effective treatment options.
* Participants must have disease that is not amenable to potentially curative resection.
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Participants with asymptomatic brain metastases and treated brain metastases are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Adequate hematological function defined by:

  * white blood cell (WBC) count greater than or equal to 3 x 10^9/L,
  * absolute neutrophil count (ANC) greater than or equal to 1.5 x10^9/L,
  * platelet count greater than or equal to 100 x 10^9/L,
  * Hemoglobin (Hgb) greater than or equal to 9 g/ dL
* Adequate hepatic function defined by:

  * a total bilirubin level less than or equal to 1.5 x upper limit of normal (ULN),
  * an aspartate aminotransferase (AST) level less than or equal to 2.5xULN, (less than or equal to 5X ULN if liver metastasis)
  * an alanine transaminase (ALT) level less than or equal to 2.5 xULN, (less than or equal to 5X ULN if liver metastasis).
* Adequate renal function defined by:

  * Creatinine OR Measured, or calculated creatinine clearance (CrCl) (estimated glomerular filtration rate (eGFR) may also be used in place of CrCl): < 1.5x institution upper limit of normal OR greater than or equal to 45 mL/min/1.73 m^2 for participant with creatinine levels greater than or equal to 1.5 X institutional ULN.

Note: Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard.

* The effects of the study treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment and up to 6 months after the last dose of the study drug (s). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Subjects must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents.
* Systemic anti-cancer treatment or major surgery within 2 weeks prior to enrollment.
* Radiotherapy within 24 hours prior to enrollment.
* Participants who require treatment with strong inhibitors or inducers of Cytochrome P450, family 3, subfamily A (CYP3A) or with uridine diphosphate glucuronosyltransferase 1A1 gene (UGT1A1) inhibitors during the planned period of investigational treatment with PLX038.
* Participants with known Gilbert's syndrome.
* Participants homozygous for the UGT1A1*28 variant allele with severely reduced UGT1A1 activity.
* Participants with known human immunodeficiency virus (HIV), hepatitis C virus (HCV), Hepatitis B virus (HBV) status on antiviral drugs are excluded due to the absence of previous experience with concurrent use of antiviral medications and the investigational drug product to be evaluated in the current study and possible for adverse pharmacokinetic and/or pharmacodynamic interactions.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PLX038 or rucaparib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that may impair the participants tolerance of study treatments.
* Pregnant women are excluded from this study because PEGSN38 and rucaparib potential for teratogenic or abortifacient effects are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PEGSN38 and rucaparib, breastfeeding should be discontinued if the mother is treated with study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0013.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The phase II portion of the study was not done because the study was closed to enrollment due to Clovis Oncology withdrawing support for the study.
Groups:
- Phase I Arm 1 Level -1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 200 mg: No participants were enrolled in this group. Phase I - Participants with solid tumors enrolled to PLX038 (PEGylated SN38) and rucaparib escalation dose levels.
  PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 200 mg by mouth (PO) PLX038: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. PLX038 (PEGylated SN38) will be administered as a 1 hour (-10 minutes / +30 minutes) intravenous (IV) infusion on Day 1 of each cycle (21 days).
  Rucaparib: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. Rucaparib will be given orally at designated dose twice a day on days 5 to 19 of every 21-day cycle.
- Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg: Phase I - Participants with solid tumors enrolled to PLX038 (PEGylated SN38) and rucaparib escalation dose levels.
  PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 400 mg by mouth (PO)
  PLX038: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. PLX038 (PEGylated SN38) will be administered as a 1 hour (-10 minutes / +30 minutes) intravenous (IV) infusion on Day 1 of each cycle (21 days).
  Rucaparib: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. Rucaparib will be given orally at designated dose twice a day on days 5 to 19 of every 21-day cycle.
- Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg: Phase I Participants with solid tumors enrolled to PLX038 (PEGylated SN38) and rucaparib escalation dose levels.
  PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 300 mg by mouth (PO)
  PLX038: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. PLX038 (PEGylated SN38) will be administered as a 1 hour (-10 minutes / +30 minutes) intravenous (IV) infusion on Day 1 of each cycle (21 days).
  Rucaparib: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. Rucaparib will be given orally at designated dose twice a day on days 5 to 19 of every 21-day cycle.
- Phase IIA Arm 2: No participants were enrolled in this group. Phase IIA Participants with small cell lung cancer (SCLC) enrolled at the maximum tolerated dose of PLX038 (PEGylated SN38) and rucaparib after the MTD of PLX038 and rucaparib is established. Level 2, PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO);Level 3, PLX038, every 3 weeks, 1.7 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO);Level 4, PLX038, every 3 weeks, 2.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO);Level 2A PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 400 mg by mouth (PO) and/or Level 3A. PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 600 mg by mouth (PO). PLX038: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. PLX038 (PEGylated SN38) will be administered as a 1hour (-10 minutes / +30 minutes) intravenous (IV) infusion on Day 1 of each cycle (21 days). Rucaparib: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. Rucaparib will be given orally at designated dose twice a day on days 5 to 19 of every 21-day cycle.
- Phase IIB Arm 2: No participants were enrolled in this group. Phase IIB Participants with extra-pulmonary small cell carcinomas enrolled at the maximum tolerated dose (MTD) of PLX038 (PEGylated SN38) and rucaparib after the MTD of PLX038 and rucaparib is established.
  Level 2, PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 3, PLX038, every 3 weeks, 1.7 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 4, PLX038, every 3 weeks, 2.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 2A PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 400 mg by mouth (PO); and/or Level 3A. PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 600 mg by mouth (PO).
  PLX038: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: MTD identified in phase I. PLX038 (PEGylated SN38) will be administered as a 1 hour (-10 minutes / +30 minutes) intravenous (IV) infusion on Day 1 of each cycle (21 days).
  Rucaparib: Phase I: Dose escalation will follow the classical 3+3 trial design by Fibonacci sequence. Phase II: Maximum tolerated dose (MTD) identified in phase I. Rucaparib will be given orally at designated dose twice a day on days 5 to 19 of every 21-day cycle.
Period: Phase I - Maximum Tolerated Dose
Arm/Group | Phase I Arm 1 Level -1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 200 mg | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg | Phase IIA Arm 2 | Phase IIB Arm 2
Started | 0 | 8 | 2 | 0 | 0
Completed | 0 | 8 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase IIA - Assess Efficacy
Arm/Group | Phase I Arm 1 Level -1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 200 mg | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg | Phase IIA Arm 2 | Phase IIB Arm 2
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase IIB - Assess Efficacy
Arm/Group | Phase I Arm 1 Level -1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 200 mg | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg | Phase IIA Arm 2 | Phase IIB Arm 2
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.06 (12.25) | 59.75 (4.17) | 57.6 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Clinical Benefit Rate
Description: Assess the efficacy with respect to clinical benefit rate (CBR) (Complete Response (CR)+ partial response (PR)+ stable disease (SD) for 4 months according to Response Evaluation Criteria (RECIST 1.1) of a combination of PLX038(PEGylated SN38) and rucaparib in previously treated participants with small cell lung cancer and extra-pulmonary small cell carcinomas. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). CR is disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Disease progression at 4 months
Population: This outcome measure was not done because the study was closed to enrollment due to Clovis Oncology withdrawing support for the study. No data was collected for this phase II outcome measure.
Arm/Group | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of PLX038 (PEGylated SN38) in Combination With Rucaparib
Description: Maximum tolerated dose (MTD) of PLX038 (PEGylated SN38) in combination with rucaparib. The MTD is the dose level at which no more than 1 of 6 participants experience dose limiting toxicity (DLT) during the DLT evaluation period, and the dose below that at which at least 2 (of 6) participants have DLT as a result of the drug. A DLT is (if deemed drug-related) a Grade 4 neutropenia that does not resolve within 7 days; Grade 4 thrombocytopenia or grade 3 thrombocytopenia complicated with hemorrhage; Grade 4 anemia that does not resolve within 7 days despite optimal therapy; Inability to begin subsequent treatment course within 21 days of the scheduled date, due to study drug toxicity.
Time Frame: One cycle, approximately 21 (+7) days
Measure: Number; unit: g/m^2
Groups:
- Phase I: All Participants: All participants who received at least one dose of PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 200 mg; PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg; and Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg.
Arm/Group | Phase I: All Participants
Number analyzed (Participants) | 10
g/m^2 | NA — MTD was not reached because dose escalation was not completed.

3. Secondary Outcome: Phase I and Phase II Grades 1-5 Serious and/or Non-serious Adverse Events Related to PLX038 (PEGylated SN38) and/or Rucaparib
Description: The safety of the treatment will be monitored, and any toxicities identified will be reported by type and grade. Toxicities were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: Date first signed consent to date off study, approximately 21 months and 18 days; and 2 months and 5 days for each group respectively.
Population: Data is reported for the phase I portion only because the study was closed to enrollment prior to phase II due to Clovis Oncology withdrawing support for the study.
Measure: Number; unit: Adverse events
Groups:
- Phase I Arm 1 Level 1 - Related to PLX038 (PEGylated SN38); Phase I - Arm 1 Level 1A - Related to PLX038 (PEGylated SN38): Phase I - Participants with solid tumors with serious and/or non-serious adverse events related to PLX038 (PEGylated SN38).
- Phase I Arm 1 Level 1 - Related to Rucaparib; Phase I - Arm 1 Level 1A - Related to Rucaparib: Phase I - Participants with solid tumors with serious and/or non-serious adverse events related to Rucaparib.
Arm/Group | Phase I Arm 1 Level 1 - Related to PLX038 (PEGylated SN38) | Phase I - Arm 1 Level 1A - Related to PLX038 (PEGylated SN38) | Phase I Arm 1 Level 1 - Related to Rucaparib | Phase I - Arm 1 Level 1A - Related to Rucaparib
Number analyzed (Participants) | 8 | 2 | 8 | 2
Adverse events
  Grade 1 Non-Serious Abdominal pain | 2 | 1 | 4 | 2
  Grade 1 Non-Serious Alanine aminotransferase increased | 0 | 0 | 3 | 0
  Grade 1 Non-Serious Alopecia | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Anemia | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Anorexia | 3 | 0 | 3 | 0
  Grade 1 Non-Serious Aspartate aminotransferase increased | 0 | 0 | 1 | 1
  Grade 1 Non-Serious Bloating | 4 | 1 | 3 | 1
  Grade 1 Non-Serious Blood bicarbonate decreased | 0 | 2 | 0 | 2
  Grade 1 Non-Serious Bruising | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Chills | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Constipation | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Diarrhea | 8 | 1 | 9 | 3
  Grade 1 Non-Serious Dysgeusia | 1 | 0 | 1 | 1
  Grade 1 Non-Serious Dysuria | 3 | 0 | 2 | 0
  Grade 1 Non-Serious Fatigue | 4 | 0 | 4 | 0
  Grade 1 Non-Serious Flatulence | 0 | 0 | 1 | 0
  Grade 1 Non-Serious Hypokalemia | 1 | 4 | 1 | 3
  Grade 1 Non-Serious Intestinal stoma site bleeding | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Lymphocyte count decreased | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Nausea | 5 | 0 | 5 | 2
  Grade 1 Non-Serious Neutrophil count decreased | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Platelet count decreased | 5 | 4 | 5 | 4
  Grade 1 Non-Serious Pruritis | 2 | 0 | 0 | 0
  Grade 1 Non-Serious Rectal hemorrhage | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Urinary frequency | 1 | 0 | 1 | 0
  Grade 1 Non-Serious Vomiting | 3 | 1 | 3 | 2
  Grade 1 Non-Serious White blood cell decreased | 2 | 1 | 2 | 1
  Grade 2 Non-Serious Abdominal pain | 3 | 0 | 6 | 0
  Grade 2 Non-Serious Alopecia | 3 | 0 | 3 | 0
  Grade 2 Non-Serious Anemia | 7 | 4 | 7 | 4
  Grade 2 Non-Serious Bloating | 2 | 0 | 3 | 1
  Grade 2 Non-Serious Diarrhea | 5 | 0 | 6 | 1
  Grade 2 Non-Serious Fatigue | 3 | 0 | 3 | 0
  Grade 2 Flatulence | 1 | 0 | 1 | 0
  Grade 2 Non-Serious Gastroesophageal reflux disease | 0 | 0 | 1 | 0
  Grade 2 Non-Serious Lymphocyte decreased | 4 | 0 | 4 | 0
  Grade 2 Non-Serious Nausea | 2 | 0 | 2 | 0
  Grade 2 Non-Serious Neutrophil count decreased | 3 | 0 | 3 | 0
  Grade 2 Non-Serious Platelet count decreased | 2 | 2 | 2 | 2
  Grade 2 Non-Serious Pruritis | 0 | 0 | 1 | 0
  Grade 2 Non-Serious Vomiting | 3 | 0 | 3 | 0
  Grade 2 Non-Serious White blood cell decreased | 2 | 0 | 2 | 0
  Grade 3 Non-Serious Abdominal pain | 0 | 0 | 1 | 0
  Grade 3 Serious Anemia | 5 | 2 | 5 | 2
  Grade 3 Serious Diarrhea | 2 | 0 | 3 | 0
  Grade 3 Serious Gastrointestinal disorders - Other specify | 0 | 1 | 0 | 1
  Grade 3 Non-Serious Lymphocyte count decreased | 4 | 1 | 4 | 1
  Grade 3 Serious Nausea | 1 | 0 | 1 | 0
  Grade 3 Non-Serious Neutrophil count decreased | 3 | 1 | 3 | 1
  Grade 3 Non-Serious Platelet count decreased | 4 | 2 | 4 | 2
  Grade 3 Serious Vomiting | 1 | 0 | 1 | 0
  Grade 3 Non-Serious White blood cell decreased | 5 | 1 | 5 | 2
  Grade 4 Serious Febrile neutropenia | 1 | 1 | 1 | 1
  Grade 4 Non-Serious Lymphocyte count decreased | 3 | 0 | 3 | 0
  Grade 4 Non-Serious Neutrophil count decreased | 1 | 1 | 1 | 1
  Grade 4 Serious Platelet Count decreased | 3 | 0 | 3 | 0
  Grade 4 Serious Sepsis | 1 | 1 | 1 | 1
  Grade 4 Non-Serious White blood cell decreased | 1 | 1 | 1 | 1
  Grade 5 Serious Gastrointestinal disorders - Other specify | 0 | 2 | 0 | 2

4. Secondary Outcome: Phase IIA Progression-free Survival (PFS)
Description: Among participants in the phase IIA cohort, median progression free survival (PFS) will be calculated from the on-study date using the Kaplan-Meier method, along with 95% confidence intervals on the median PFS. PFS is defined as the time from on-study date to documented evidence of disease progression. Disease progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And appearance of one or more new lesions.
Time Frame: Time from the on-study date to documented evidence of disease progression
Population: This outcome measure was not done because the study was closed to enrollment due to Clovis Oncology withdrawing support for the study. No data was collected for this phase IIA outcome measure.
Groups:
- Phase IIA Arm 2: Phase IIA Participants with small cell lung cancer (SCLC) enrolled at the maximum tolerated dose (MTD) of PLX038 (PEG~SN-38) and rucaparib after the MTD of PLX038 and rucaparib is established.
  Level 2, PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 3, PLX038, every 3 weeks, 1.7 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 4, PLX038, every 3 weeks, 2.3 g/m^2, intravenous (IV); Rucaparib, days 3-19 twice a day (BID), total dose, 600 mg by mouth (PO); Level 2A PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 400 mg by mouth (PO); and/or Level 3A. PLX038, every 3 weeks, 1.3 g/m^2, intravenous (IV); Rucaparib, days 5-19 twice a day (BID), total dose, 600 mg by mouth (PO).
Arm/Group | Phase IIA Arm 2
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase IIA Overall Survival
Description: Among participants in the phase IIA cohort, median overall survival (OS) will be calculated from the on-study date using the Kaplan-Meier method, along with 95% confidence intervals on the median OS.OS is defined as the date of on-study to the date of death from any cause or last follow-up.
Time Frame: Date of on-study to the date of death from any cause or last follow-up
Population: as for outcome 4
Arm/Group | Phase IIA Arm 2
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase I - Number of Participants Who Experience a Clinical Response (Complete Response (CR)+Partial Response (PR)
Description: The number of participants who experience a clinical response (Complete Response (CR)+Partial Response (PR) will be reported. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). CR is disappearance of all target lesions; any pathological lymph nodes must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Disease progression, a median of 43 days with range of 20 to 350 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg
Number analyzed (Participants) | 8 | 2
Participants
  Complete Response | 1 | 0
  Partial Response | 1 | 0

7. Other Pre Specified Outcome: Phase I Number of Participants With a Dose Limiting Toxicity (DLT)
Description: A DLT is (if deemed drug-related) Grade 4 neutropenia that does not resolve within 7 days; Grade 4 thrombocytopenia or grade 3 thrombocytopenia complicated with hemorrhage; Grade 4 anemia that does not resolve within 7 days despite optimal therapy; Inability to begin subsequent treatment course within 21 days of the scheduled date, due to study drug toxicity.
Time Frame: One cycle, approximately 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg
Number analyzed (Participants) | 8 | 2
Participants | 1 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg
Number analyzed (Participants) | 8 | 2
Participants | 8 | 2

ADVERSE EVENTS:
Time Frame: Date first signed consent to date off study, approximately 21 months and 18 days; and 2 months and 5 days for each group respectively.
Arm/Group | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg
All-Cause Mortality (participants affected / at risk) | 7/8 | 2/2
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/2
Other Adverse Events (participants affected / at risk) | 8/8 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg (N=8) | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, Neutropenic Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Injury, poisoning and procedural complications - Other, Traumatic Head Injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Arm 1 Level 1, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 400 mg (N=8) | Phase I - Arm 1 Level 1A, PLX038 (PEGylated SN38) 1.3 g/m^2 and Rucaparib 300 mg (N=2)
Abdominal pain (Gastrointestinal disorders) | 5 (11) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (12) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 4 (7) | 2 (2)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain - cardiac (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (17) | 2 (4)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 6 (8) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4) | 2 (6)
Hypokalemia (Metabolism and nutrition disorders) | 5 (12) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (8) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Injury, poisoning and procedural complications - Other, Traumatic Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (12) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (8) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 5 (13) | 2 (8)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (7) | 2 (2)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 5 (10) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT04209595/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04209595/ICF_001.pdf